CLINICAL TRIAL: NCT06538831
Title: A 2x2 Factorial Randomized Controlled Trial to Elucidate How Ultra-processed Foods Modulate Cardiometabolic Risk
Brief Title: Impact of Ultra-processed Foods on Cardiometabolic Risk Factors
Acronym: NOVA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Benoit Lamarche, Study director, Laval University
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NUTRISS-NOVA-2024-219
Record Dates: First submitted 2024-07-31; First posted 2024-08-06 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Cardiometabolic Risk

STUDY DESIGN:
Intervention Model Description: Parallel group 2x2 factorial randomized controlled trial in fully controlled feeding conditions
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Diet N-P- (Experimental)
  Interventions: Other: Diet N-P-
- Diet N+P- (Experimental)
  Interventions: Other: Diet N+P-
- Diet N-P+ (Experimental)
  Interventions: Other: Diet N-P+
- Diet N+P+ (Experimental)
  Interventions: Other: Diet N+P+

INTERVENTIONS:
Other: Diet N-P- — Low in saturated fatty acids (SFAs), free sugar and sodium; Low in ultra-processed foods (UPFs)
  Arms: Diet N-P-
Other: Diet N+P- — Rich in SFAs, free sugar and sodium; Low in UPFs
  Arms: Diet N+P-
Other: Diet N-P+ — Low in SFAs, free sugar and sodium; High in UPFs
  Arms: Diet N-P+
Other: Diet N+P+ — Rich in SFAs, free sugar and sodium; High in UPFs
  Arms: Diet N+P+

SUMMARY:
The goal of this clinical trial is to examine in a 2x2 factorial RCT what feature(s) of ultra-processed foods (UPFs) contribute to cardiometabolic risk in men and women. The project's hypotheses are :

1. that the nutrient composition of UPFs (high SFA, free sugar and sodium) per se has deleterious impacts on cardiometabolic risk factors;
2. that the industrial techniques and processes of UPFs per se do not.

Participants will be randomly assigned to one of 4 groups consistent with the 2x2 factorial design of the study: 1- the nutrient composition of foods (low vs. high in SFA, free sugar and sodium) and 2- the degree of industrial techniques and food processing (little to no vs.important amounts of UPFs). All foods will be provided to participants under isocaloric conditions during the 6-week dietary intervention. Participants will have to consume one of the 4 experimental diets for 6 weeks.

DETAILED DESCRIPTION:
This study is a parallel group 2x2 factorial randomized controlled trial, in which diet is fully controlled. A total of 120 men and women covering a broad range of adiposity and cardiometabolic risk factors will be randomly assigned to one of four 6-week experimental diets:

1. A diet low in saturated fatty acids (SFAs), free sugar and sodium, with low ultra-processed foods (UPFs)
2. A diet rich in SFAs, free sugar and sodium, with low UPFs;
3. A diet low in SFAs, free sugar and sodium, with high levels of UPFs;
4. A diet rich in SFAs, free sugar and sodium, with high levels of UPFs.

All foods in this full-feeding trial will be managed or prepared by food technicians at the Clinical Investigation Unit of our research center. A cyclic seven-day menu plan will be developed with similar foods across the four diets. Classifications of the degree of food processing will be made using NOVA classification. NOVA identifies four categories of foods based on the degree of food processing: 1- Unprocessed or minimally processed foods, 2- Processed Culinary Ingredients, 3- Processed Food and 4- Ultra-processed foods (UPFs). The two diets high in UPFs will predominantly feature commercially-bought foods classified as NOVA-4, while the two diets low in UPFs diets will predominantly include foods prepared in our metabolic kitchen (NOVA 1 to 3). Diets will be provided under isocaloric conditions to maintain body weight constant. The breakfast meal will represent approximately 30% of the daily energy intake in each diet, whereas the lunch and dinner meals each will provide about 35% of daily energy intake. Participants will have to come to the research center 3 to 5 times a week during the 6-week intervention to collect their meals and be weighed. Primary and secondary outcomes will be measured at the beginning and at the end of the 6-wk diet intervention.

The specifics objectives of this 2x2 factorial RCT are:

Obj 1: To assess the impact of the nutrient composition of UPFs on cardiometabolic risk, independent of variations in industrial techniques and processes (factor 1).

Obj 2: To assess the impact of industrial techniques and processes of UPFs on cardiometabolic risk, independent of variations in nutrient composition (factor 2).

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI):18 to 35 kg/m2
* Stable weight over the last 3 months (variation of less than 5 kg)
* LDL-cholesterol < 5.0 mmol/L
* HbA1c < 6.5%
* Office blood pressure <150/90 mmHg
* Non-smokers or smokers of less than 10 cigarettes a day

Exclusion Criteria:

* Pregnant or breast-feeding women
* Alcohol consumption of more than 7 drinks per week
* Women: contraceptives for less than 3 months or hormone therapy for less than 6 months
* Medication to treat hypercholesterolemia, diabetes or hypertension
* Diagnosis of cardiovascular disease, diabetes, hypertension, cancer
* Food allergies or aversions to any of the foods on the experimental menus
* Being on a diet or following a special diet
* Daytime MAPA blood pressure >150/90

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-09-25 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Post treatment fasting LDL-C concentrations | 6 weeks
  Fasting serum LDL-C concentrations (mmol/L) will be measured at the end of the 6-wk intervention in all subjects in each group, on two consecutive days post-treatment. The mean of the two post-treatment values will be used in the analyses. Analyses will be adjusted for LDL-C concentrations values measured at baseline.
Post treatment insulin sensitivity (HOMA-IR) | 6 weeks
  Insulin sensitivity (HOMA-IR) will be measured in the fasted state at the end of the 6-wk intervention in all subjects in each group, on two consecutive days post-treatment. The mean of the two post-treatment values will be used in the analyses. Analyses will be adjusted for insulin sensitivity (HOMA-IR) values measured in the fasted state at baseline.
Post treatment day-time ambulatory systolic blood pressure | 6 weeks
  Day-time ambulatory systolic blood pressure will be measured at the end of the 6-wk intervention in all subjects in each group. Analyses will be adjusted for day-time ambulatory systolic blood pressure values measured at baseline.

SECONDARY OUTCOMES:
Post treatment fasting triglyceride | 6 weeks
  Fasting serum triglyceride (mmol/L) will be measured at the end of the 6-wk intervention in all subjects in each group, on two consecutive days post-treatment. The mean of the two post-treatment values will be used in the analyses. Analyses will be adjusted for triglyceride concentrations values measured at baseline.
Post treatment ApoB-100 | 6 weeks
  Fasting serum ApoB-100 (mmol/L) will be measured at the end of the 6-wk intervention in all subjects in each group, on two consecutive days post-treatment. The mean of the two post-treatment values will be used in the analyses. Analyses will be adjusted for ApoB-100 concentrations values measured at baseline.
Post treatment HDL-C concentrations | 6 weeks
  Fasting serum HDL-C concentrations (mmol/L) will be measured at the end of the 6-wk intervention in all subjects in each group, on two consecutive days post-treatment. The mean of the two post-treatment values will be used in the analyses. Analyses will be adjusted for HDL-C concentrations values measured at baseline.
Post treatment fasting glucose concentrations | 6 weeks
  Fasting serum glucose concentrations (mmol/L) will be measured at the end of the 6-wk intervention in all subjects in each group, on two consecutive days post-treatment. The mean of the two post-treatment values will be used in the analyses. Analyses will be adjusted for glucose concentrations values measured at baseline.
Post treatment fasting insulin concentrations | 6 weeks
  Fasting serum insulin concentrations (mmol/L) will be measured at the end of the 6-wk intervention in all subjects in each group, on two consecutive days post-treatment. The mean of the two post-treatment values will be used in the analyses. Analyses will be adjusted for insulin concentrations values measured at baseline.
Post treatment day-time ambulatory diastolic blood pressure | 6 weeks
  Day-time ambulatory diastolic blood pressure will be measured at the end of the 6-wk intervention in all subjects in each group. Analyses will be adjusted for day-time ambulatory diastolic blood pressure values measured at baseline.
Post treatment 24-hr ambulatory systolic blood pressure | 6 weeks
  24-hr ambulatory systolic blood pressure will be measured at the end of the 6-wk intervention in all subjects in each group. Analyses will be adjusted for 24-hr ambulatory systolic blood pressure values measured at baseline.
Post treatment 24-hr ambulatory diastolic blood pressure | 6 weeks
  24-hr ambulatory diastolic blood pressure will be measured at the end of the 6-wk intervention in all subjects in each group. Analyses will be adjusted for 24-hr ambulatory diastolic blood pressure values measured at baseline.
On-treatment Diet palatability | 6 weeks
  These are exploratory analyses. Scales measuring diet palatability will be completed during the same three days of the 7-day cycling menu during the first and last week of the 6-wk intervention. The mean of all measurements will be used in the analyses. Title of the scale: Main course evaluation.
  Minimum and maximum values : 1 to 8 . Higher scores are not synonymous of better or worse results.
On-treatment Perceived healthiness of meals | 6 weeks
  These are exploratory analyses. Scales measuring perceived healthiness of meals will be completed during the same three days of the 7-day cycling menu during the first and last week of the 6-wk intervention. The mean of all measurements will be used in the analyses. Title of the scale: Opinion on your main course. Minimum and maximum values : 1 to 8 . Higher scores are not synonymous of better or worse results.
On-treatment Hunger and fullness perceptions | 6 weeks
  These are exploratory analyses. Scales measuring hunger and fullness perceptions will be completed during the same three days of the 7-day cycling menu during the first and last week of the 6-wk intervention. The mean of all measurements will be used in the analyses.
  Title of the scale: Visual Analogue Scale - How hungry do you feel? Minimum and maximum values : Not hungry at all to very hungry. Higher scores are not synonymous with better or worse results.
  Title of the scale: Visual Analogue Scale - How full do you feel? Minimum and maximum values : Not at all full to very full. Higher scores are not synonymous of better or worse results.
Post-treatment Gut microbiota | 6 weeks
  These are exploratory analyses in a subset of participants only. Deep 16S rDNA metagenomic analysis in feces collected at week 6 will be used to characterize gut microbiota composition and function. Analyses will be adjusted for baseline values of gut microbiota composition and function measured on fecal samples collected at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Benoît Lamarche, PhD, Principal Investigator — Laval University
Locations (1):
- Centre Nutrition, santé et société (NUTRISS), INAF, Université Laval, Québec, Quebec, Canada